CLINICAL TRIAL: NCT03467867
Title: A Phase II Study of Venetoclax and Rituximab/Hyaluronidase Human in Relapsed/Refractory CLL
Brief Title: A Study of Venetoclax and Rituximab/Hyaluronidase Human in Relapsed/Refractory CLL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1502
Record Dates: First submitted 2018-03-12; First posted 2018-03-16 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Leukemia; Venetoclax; Rituximab; Lymphoid; Lymphoproliferative Disorders; Antineoplastic Agents; Neoplasm
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Lymphoproliferative Disorders; Neoplasms | interventions — venetoclax; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venetoclax + Rituximab (Experimental): Participants will be initially placed in a venetoclax 5 weeks ramp-up period, and will be administered an initial 20 mg oral tablet dose once daily (QD), incrementing weekly up to a maximum dose of 400 mg. Participants will then continue taking venetoclax 400 mg QD from Week 5 onwards, as directed by the investigator in combination with rituximab 375 mg/m^2 IV on Day 1 of Cycle 1 followed by 13.4 mL of rituximab SC 1,600 mg/26,800 Units vial (1,600 mg rituximab and 26,800 Units hyaluronidase human) on Day 1 of Cycle 2-6.
  Interventions: Drug: Venetoclax; Drug: Rituximab; Drug: Rituximab/Hyaluronidase Human

INTERVENTIONS:
Drug: Venetoclax — Venetoclax will be administered as described in the reporting arm.
  Other Names: GDC-0199; ABT-199
Drug: Rituximab — Rituximab (IV) will be administered as described in the reporting arm.
  Other Names: Rituxan
Drug: Rituximab/Hyaluronidase Human — Rituximab/Hyaluronidase Human (SC) ill be administered as described in the reporting arm.
  Other Names: Rituxan Hycela

SUMMARY:
This is an open-label, multicenter, Phase II study to investigate the efficacy and safety of venetoclax in combination with Rituximab/hyaluronidase human in participants with relapsed or refractory chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
The study has one arm and all the patients will receive venetoclax and rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Ability and willingness to comply with the requirements of the study protocol
* Patient must have diagnosis of CLL that meets published 2008 IWCLL NCI-WG criteria.
* Patient must have relapsed/refractory disease with an indication for treatment.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2
* Adequate hematologic function (unless caused by underlying disease, as established by extensive bone marrow involvement or as a result of hypersplenism secondary to the involvement of the spleen by lymphoma per the investigator) defined as follows:

  * Hemoglobin (> / =) 9 g/dL
  * Absolute neutrophil count (> / =) 1.0 x 109/L
  * Platelet count (> / =)75 x 109/L
* Adequate renal function, as indicated by:

  * Calculated creatinine clearance ≥ 30 mL/min using 24-hour Creatinine Clearance or modified Cockcroft-Gault equation (eCCR; with the use of ideal body mass [IBM] instead of mass)
* Adequate liver function, as indicated by:

  * AST or ALT (< / =) 2.5 x ULN
  * Total bilirubin < 1.5 x ULN (or (< / =) 3 x ULN for patients with documented Gilbert syndrome)
* Female patients who are not of child-bearing potential and female patients of child-bearing potential who have a negative serum pregnancy test within 3 days prior to Cycle 1, Day 1.
* Patients with HIV infection could be included in the study, as long as their disease is under control on anti-retroviral therapy. Precautions should be taken to modify their HAART regimen to minimize drug interaction
* Warfarin is considered a cautionary medication. Patients on warfarin will be encouraged to replace warfarin with other anticoagulants if possible. If it is not possible or patient is not willing to switch, they could still be included in the study with caution.

Exclusion Criteria:

* Known hypersensitivity to any of the study drugs
* Allogeneic stem cell transplant within the past 1 year.
* Richter's transformation confirmed by biopsy
* History of other malignancy that could affect compliance with the protocol or interpretation of results

  * Patients with a history of curatively treated basal or squamous cell carcinoma or Stage 1 melanoma of the skin or in situ carcinoma of the cervix are eligible.
  * Patients with a malignancy that has been treated with surgery alone with curative intent will be included. Individuals in documented remission without treatment for (> / =) 2 years prior to enrollment may be included at the discretion of the investigator.
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results or that could increase risk to the patient, including renal disease that would preclude chemotherapy administration or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1, Day 1
* Received the following agents within 7 days prior to the first dose of venetoclax:

  * Steroid therapy for anti-neoplastic intent
  * Strong and moderate CYP3A inhibitors
  * Strong and moderate CYP3A inducers
  * Consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or star fruit within 3 days prior to the first dose of venetoclax
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Presence of positive test results for hepatitis B virus (HBV), hepatitis B surface antigen (HBsAg), or hepatitis C (HCV) antibody
* Patients who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation
* Patients with occult or prior HBV infection (defined as positive total hepatitis B core antibody [HBcAb] and negative HBsAg) may be included if HBV DNA is undetectable. These patients must be willing to undergo monthly DNA testing.
* Known infection with human T-cell leukemia virus 1 (HTLV-1)
* Patients with uncontrolled HIV infection
* Receipt of live-virus vaccines within 28 days prior to the initiation of study treatment or need for live-virus vaccines at any time during study treatment
* Pregnant or lactating, or intending to become pregnant during the study Women of childbearing potential must have a negative serum pregnancy test result within 21 days prior to initiation of study drug.
* Recent major surgery (within 6 weeks prior to the start of Cycle 1, Day 1) other than for diagnosis
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Known allergy to both xanthine oxidase inhibitors and rasburicase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Baseline up to disease progression or death, whichever occurs first (up to approximately 5 years)
  Percentage of Participants With Best Overall Response (OR)(Defined as Complete Response [CR], Initial CR [CRi], Nodular Partial Response [nPR], PR) as Assessed by Investigator Determined Using iwCLL Guidelines

SECONDARY OUTCOMES:
Disease Response | 12 weeks after Day 1 of last cycle of combination therapy (approximately 5 years, cycle length= 28 days)
  Percentage of Participants With Disease Response (OR, CR, CRi, nPR, PR) as Assessed by Investigator Determined Using iwCLL Guidelines at end of Combination Treatment Visit
Duration of Responses (DOR) | Baseline up to disease progression or death, whichever occurs first (up to approximately 5 years)
  Duration of Responses (DOR)
Time to Progression (TTP) | Baseline up to disease progression or death, whichever occurs first (up to approximately 5 years)
  Time to progression will be defined as the time from the date of first dose (date of enrollment if not dosed) to the date of earliest disease progression (per the investigator assessment).
Progression-Free Survival (PFS) | Baseline up to disease progression or death, whichever occurs first (up to approximately 5 years) ]
  Investigator-Assessed Progression-Free Survival (PFS) Determined Using Standard International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Guidelines
Overall Survival (OS) | Baseline up to death (up to approximately 5 years)
  Overall Survival (OS)
Time to Next Anti-CLL Treatment (TTNT) | Baseline up to disease progression or death, whichever occurs first (up to approximately 5 years) ]
  Time to Next Anti-CLL Treatment (TTNT)
Percentage of Participants With Minimal Residual Disease (MRD) | 12 weeks after Day 1 of last cycle of combination therapy (up to approximately 5 years, cycle length= 28 days) ]
  Percentage of Participants With Minimal Residual Disease (MRD) Negativity at End of Combination Treatment Response Visit

CONTACTS AND LOCATIONS:
Overall Officials: Kieron Dunleavy, MD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey